CLINICAL TRIAL: NCT05591898
Title: The Effect of Progressive Relaxation Exercises on Preoperative Anxiety and Postoperative Pain in Bariatric Surgery Patients
Brief Title: The Effect of Progressive Relaxation Exercises on Bariatric Surgery Period
Acronym: PREbari
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Atlas University (Other); Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ismail Calikoglu, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAEK/2022.01.7
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Anxiety; Postoperative Pain
Keywords: bariatric surgery; Progressive relaxation exercises; anxiety; postoperative pain
MeSH Terms: conditions — Obesity, Morbid; Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercises group (Experimental): Participants will be randomly selected by a computer based system (Block randomization was used to keep the sample size of the groups similar. Random Allocation Software (Ver. 1.0.0) will be used to allocate the patients to groups). Selected participants will be invited to a meeting which will be held face-to-face and in a quiet environment. Progressive Relaxation Exercises will be explained to this group in a step-by-step manner whose surgery date is determined to undergo bariatric surgery by the relevant researcher. After this stage, participants will be followed to do the exercises regularly for a month by a researcher. Patients will fill the Amsterdam Preoperative Anxiety and Information Score Scale preoperatively at the hospital. After the surgery, the patients will be evaluated by the researchers in terms of pain scores and analgesic usage frequency in the recovery room and 1st, 4th, 8th, 12th, 24th, 36th and 48th hours data will be collected in the postoperative service.
  Interventions: Behavioral: Progressive relaxation exercises
- Control group (No Intervention): This group will be the randomized selected patients who will not get any intervention. Patients will fill the Amsterdam Preoperative Anxiety and Information Score Scale preoperatively at the hospital. After the surgery, the patients will be evaluated by the researchers in terms of pain scores and analgesic usage frequency in the recovery room and 1st, 4th, 8th, 12th, 24th, 36th and 48th hours data will be collected in the postoperative service.

INTERVENTIONS:
Behavioral: Progressive relaxation exercises — Training booklet and CD as a guide on the implementation of Progressive Relaxation Exercises prepared by the Turkish Psychological Association; muscle relaxation exercises, rhythmic breathing and music recital. In the first 10 minutes of this three-part CD, the definition and purpose of deep relaxation and the practices to be considered during exercise are explained. In the second part of 30 minutes; relaxation exercises are explained with the sound of the stream and verbal instructions. The third part, consisting of 30 minutes; it contains only relaxation music without instructions.
  Arms: Progressive relaxation exercises group

SUMMARY:
The goal of this clinical trial is to test the effect of the progressive relaxation exercises in perioperative bariatric surgery patient care. The investigators know that the preoperative anxiety is an important factor that affects acute postoperative pain experience. Additionally, the investigators know that there is a relationship between preoperative anxiety and moderate to severe pain in the first 12 hours postoperatively, and this is also true for patients undergoing bariatric surgery. The main questions it aims to answer are:

* Does preoperative anxiety level of patient who will undergo bariatric surgery and who are applied progressive relaxation exercises is lower than those who did not apply exercise?
* Does postoperative pain level of patient who underwent bariatric surgery and applied progressive relaxation exercises was lower than patients who did not apply exercise?

Participants will be randomly split into two groups and one of the groups of participants will learn how to do progressive relaxation exercises preoperatively and the other group will learn nothing. Then at the time of the surgery, all participants will fill a survey preoperatively to analyze participants' anxiety level in each group and the investigators will collect data about participants' pain level postoperatively.

Researchers will compare these data whether there is an effect of the progressive relaxation exercises on preoperative anxiety and postoperative pain or not.

DETAILED DESCRIPTION:
Preoperative anxiety is a defined factor that affects the acute postoperative pain experience. There is an evidence-based relationship between preoperative anxiety and moderate to severe pain in the first 12 hours postoperatively. Similarly, patients with high anxiety before bariatric surgery experienced more pain in the first postoperative hour. Interventions to reduce anxiety may decrease the surgical pain response and improve postoperative recovery by reducing the sympathetic nervous system response. There are various pharmacological and non-pharmacological methods (such as education, music, acupuncture, massage) used for preoperative anxiety. One of the non-pharmacological methods is progressive relaxation exercises. Progressive muscle relaxation is a relaxation technique developed by Edmund Jacobson in the 1920s. It is one of the simple and easy to learn relaxation techniques. These exercises involve contracting muscles to create tension and gradually releasing that tension. It is routinely repeated until complete relief is achieved. In the literature, there are studies on the effect of progressive relaxation exercises on anxiety and pain. In these studies, it was determined that progressive relaxation exercises reduce anxiety, pain, muscle tension, sleep disorders and fatigue levels. No study has been found on the effect of progressive relaxation exercises on preoperative anxiety and postoperative pain in bariatric surgery patients.

So, the investigators planned a study to determine the effect of progressive relaxation exercises on preoperative anxiety and postoperative pain in patients undergoing bariatric surgery.

Patients willing to have a bariatric surgery in our hospital will be split into two groups randomly and one of the groups of participants will be learnt how to do progressive relaxation exercises one month preoperatively and the other group will learn nothing. Then at the time of the surgery, all patients will fill a survey preoperatively to collect the participants' anxiety level in each group and pain scores will be collected postoperatively. All patients will give informed consent to join to the study.

H1: Preoperative anxiety level of patients who will undergo bariatric surgery and who are applied progressive relaxation exercises is lower than those who do not exercise.

H2: Postoperative pain level of patients who underwent bariatric surgery and applied progressive relaxation exercises was lower than patients who did not apply exercise.

Study arms are explained below.

ELIGIBILITY:
Inclusion Criteria:

* Having bariatric surgery plan (such as sleeve gastrectomy, gastric bypass),
* 18 years and over,
* Do not have any medically diagnosed health problems (neurological, psychiatric, orthopedic) that will prevent learning and practicing progressive muscle relaxation exercises,
* Agreeing to apply progressive relaxation exercises, willing and willing to participate in the study,
* Patients who do not know and practice progressive relaxation exercises before will be included in the study.

Exclusion Criteria:

* Patients younger than 18 and older than 65,
* Patients who do not want to apply progressive relaxation exercises,
* who do not apply them as desired during the study period,
* who have health problems (neurological, psychiatric, orthopedic) that may affect their ability to do the exercises will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety level | Preoperatively
  The Progressive relaxation exercises supposed to lower the preoperative anxiety level in bariatric surgery patients. The patients will fill the Amsterdam Preoperative Anxiety and Information Score Scale preoperatively. The Amsterdam Preoperative Anxiety and Information Scale is a self-report questionnaire composed of six questions that were developed and validated to evaluate a patient's preoperative anxiety. The range of the scale is between 6 to 30 and higher means more anxiety.

SECONDARY OUTCOMES:
Postoperative pain level | Postoperative pain scores collection is planned at the postoperative period in the first 48 hour after the surgery.
  Progressive relaxation exercises supposed to lower the postoperative pain scores in the bariatric surgery patients. The pain score will be identified by using the visual analog scale (VAS) score. VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The range of the scale is between 0 to 10 and higher means more pain.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Çalıkoğlu, M.D., Principal Investigator — Başakşehir Çam & Sakura Şehir Hospital; İsmail Çalıkoğlu, Study Director — Başakşehir Çam & Sakura Şehir Hospital
Locations (1):
- Başakşehir Çam & Sakura Şehir Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the study will be reported as an article in a high quality journal.

REFERENCES:
- [Background] Daniel S, Sindhu JV. Effectiveness of Progressive Muscle Relaxation Technique on Post Operative Pain and Anxiety Among patients Who Have Undergone Abdominal Surgery. International Journal of Nursing Critical Care. 2020; 6(1), 35-41.
- [Background] David LA, Sijercic I, Cassin SE. Preoperative and post-operative psychosocial interventions for bariatric surgery patients: A systematic review. Obes Rev. 2020 Apr;21(4):e12926. doi: 10.1111/obr.12926. Epub 2020 Jan 22. PMID 31970925
- [Background] Felix MMDS, Ferreira MBG, Oliveira LF, Barichello E, Pires PDS, Barbosa MH. Guided imagery relaxation therapy on preoperative anxiety: a randomized clinical trial. Rev Lat Am Enfermagem. 2018 Nov 29;26:e3101. doi: 10.1590/1518-8345.2850.3101. PMID 30517586
- [Background] Gravani S, Matiatou M, Nikolaidis PT, Menenakos E, Zografos CG, Zografos G, Albanopoulos K. Anxiety and Depression Affect Early Postoperative Pain Dimensions after Bariatric Surgery. J Clin Med. 2020 Dec 25;10(1):53. doi: 10.3390/jcm10010053. PMID 33375765
- [Result] Alvarez-Garcia C, Yaban ZS. The effects of preoperative guided imagery interventions on preoperative anxiety and postoperative pain: A meta-analysis. Complement Ther Clin Pract. 2020 Feb;38:101077. doi: 10.1016/j.ctcp.2019.101077. Epub 2019 Dec 4. PMID 32056813